CLINICAL TRIAL: NCT06095453
Title: Evaluation of the Analgesic Efficacy of Multimodal Pain Control Regimens That Aim to Limit the Use of Narcotics in Cholecystectomy and Hernia Repairs
Status: Active, not recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 124.SUR.2022.M
Record Dates: First submitted 2023-07-06; First posted 2023-10-23 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Narcotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Pain control regimens — Narcotics in cholecystectomy and hernia repairs
  Other Names: Narcotics

SUMMARY:
Subjects were patients of the five surgeons with Surgical Associates of Mansfield (SAM) who underwent an elective or urgent laparoscopic cholecystectomy; or elective or urgent laparoscopic or open hernia repair (inguinal, ventral, or umbilical); and who otherwise met the inclusion criteria. I

DETAILED DESCRIPTION:
This performance improvement study is a retrospective review of data obtained from patients at Methodist Mansfield Medical Center (MMMC) in Mansfield, Texas from May 1, 2022 to September 30, 2022. Subjects were patients of the five surgeons with Surgical Associates of Mansfield (SAM) who underwent an elective or urgent laparoscopic cholecystectomy; or elective or urgent laparoscopic or open hernia repair (inguinal, ventral, or umbilical); and who otherwise met the inclusion criteria. Incisional hernias were excluded. Emergent hernia operations that required bowel or colon resections due to strangulation were excluded

ELIGIBILITY:
Inclusion Criteria:

Patients of the five physicians of the SAM group Patients ≥18 years Patients undergoing urgent or elective laparoscopic and robotic cholecystectomy OR patients undergoing urgent or elective laparoscopic, robotic or open hernia repair (ventral, umbilical, or inguinal).

Exclusion Criteria:

Patients <18 years Patients with chronic pain conditions managed with chronic use of narcotics Patients that underwent incisional hernia repairs Patients that underwent complicated hernia repairs that included other operations such as colon and bowel resection procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects were patients of the five surgeons with Surgical Associates of Mansfield (SAM) who underwent an elective or urgent laparoscopic cholecystectomy; or elective or urgent laparoscopic or open hernia repair (inguinal, ventral, or umbilical); and who otherwise met the inclusion criteria. Incisional hernias were excluded. Emergent hernia operations that required bowel or colon resections due to strangulation were excluded
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Narcotics Doses and timeframe | 4 months
  number of doses of narcotics taken including the number of times refilled.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Trussell, MD, Principal Investigator — Mansfield
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
8.5. Data Use and Sharing Study data or any protected health information will not be shared with anyone that is not delegated to the study. The PI is committed to disseminate research results in a timely fashion. Sharing of results generated by the data analysis during the course of the project will be through presentation at national scientific meetings and/or publication in open access journals. All information obtained will be source de-identified and presented on a large scale and not traceable to any one particular individual.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: Medical Electronic devices